CLINICAL TRIAL: NCT06315010
Title: A Phase II Study Assessing Safety and Efficacy of REPotrectinib in ROS1-positive Non-small Cell Lung Cancer Patients With Active Brain mEtastasis (REPOSE Study)
Brief Title: REPotrectinib in ROS1-positive Non-small Cell Lung Cancer Patients With Active Brain mEtastasis
Acronym: REPOSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP662; 2023-508112-35-00 (EU CTIS Number); CA127-1061 (Other: Bristol-Myers Squibb GmbH & Co)
Record Dates: First submitted 2024-02-16; First posted 2024-03-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: NSCLC; Brain Metastases; ROS1 Gene Rearrangement
Keywords: Metastatic NSCLC; Brain metastasis; ROS1; Repotrectinib
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — repotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repotrectinib (Experimental): Repotrectinib 160 mg orally (PO) every day (QD) for 14 days, and 160 mg twice a day (BID) thereafter.
  Interventions: Drug: Repotrectinib

INTERVENTIONS:
Drug: Repotrectinib — Repotrectinib is administered orally in capsule form, with each capsule containing size 0 hard gelatin 40 mg of the active compound in bottles containing 30 capsules.
  Repotrectinib is administered orally in the form of capsules. The capsules are taken by mouth and swallowed intact (without chewing, crushing, or opening) with water or another suitable liquid.
  Other Names: BMS-986472; TPX-0005

SUMMARY:
REPOSE is a phase II clinical trial exploring the safety and efficacy of repotrectinib in patients with non-small cell lung cancer (NSCLC) characterized by the presence of brain metastasis (BM) and whose tumors have mutated ROS proto-oncogene 1, receptor tyrosine kinase (ROS1) gene.

DETAILED DESCRIPTION:
REPOSE is an international multicenter, open-label, single arm phase II clinical trial designed to evaluate the efficacy of repotrectinib in patients with ROS1-positive NSCLC with BM.

Upon meeting all selection criteria, a total of 20 participants confirmed ROS1 rearrangement will be enrolled. Participants who have received prior chemotherapy, immunotherapy or other non-ROS1 tyrosine kinase inhibitor (TKI) are eligible.

Patients will continue study treatment until end of treatment (EoT) defined as the date of disease progression, death, or discontinuation from the study treatment for any other reason. After study treatment discontinuation, all participants will undergo a safety visit (at 28 ± 7 days after last treatment dose) in order to follow up toxicities and changes in concomitant medication. Patients discontinuing the study treatment at any time will enter a post-treatment follow-up period during which survival and subsequent anticancer therapy information will be collected every 3 months (± 7 days) from the safety visit until death, lost to follow-up, elective withdrawal from the study, or the end of study (EoS), whichever occurs first. Patients who discontinue treatment without evidence of disease progression will be also followed for tumor assessments until documented progression, elective withdrawal from the study, the start of new anti-cancer treatment, or the EoS.

EoS is estimated to occur approximately 13 months after the last patient included in the study initiates repotrectinib treatment, unless consent withdrawal, patient is lost to follow-up, death, or premature termination of the study. EoS is defined as the last data collection point at the last participant's safety visit and will occur after the study treatment termination of the last patient in the study.

The main objective of REPOSE study is to determine the efficacy of repotrectinib at any timepoint during the study period as determined locally by best central nervous system (CNS) response, that is in terms of intracranial objective response rate (IC-ORR).

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study only if they meet all the following criteria:

1. Patient must be capable to understand the purpose of the study and have signed written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female or male patients ≥ 18 years of age at the time of signing ICF.
3. Patients must be capable to swallow capsules intact (without chewing, crushing, or opening).
4. Histologically documented NSCLC.
5. Patients may have active brain metastases with or without related symptoms.
6. No indication for immediate local therapy (neurosurgery, brain radiotherapy) of brain metastases per local investigator.

   Note: in case of immediate local therapy is needed, the study's medical monitor should be consulted.
7. Type II leptomeningeal disease per European Association of Neuro-Oncology (EANO) - European Society for Medical Oncology (ESMO) Clinical Practice Guidelines are allowed.
8. Patients with confirmed ROS1 rearrangement. Prior to study enrollment, patients must have had confirmation of ROS1 rearrangement, which should have been determined locally by a certified laboratory using methods such as fluorescent in situ hybridization (FISH), next generation sequencing (NGS), quantitative PCR (qPCR), or immunohistochemistry (IHC).
9. Measurable disease according to RANO-BM criteria, with at least one measurable brain lesion of ≥10 mm on T1-weighted, gadolinium-enhanced magnetic resonance imaging (MRI).
10. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
11. Minimum life expectancy of ≥ 6 weeks at screening.
12. No limit in number of prior chemotherapies, immunotherapy or other non-ROS1 TKI regimens. De novo patients can also be included.
13. Patients must not have previously received any ROS1 TKI-based treatment.
14. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
15. If feasible, archival tumor biopsy sample at baseline (from primary tissue or any metastatic site) should be provided.
16. Patient has adequate bone marrow, liver, and renal function:

    I. Hematological (without platelet, red blood cell transfusion, and/or granulocyte colony-stimulating factor support within 28 days before first study treatment dose): White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 8.0 g/dL (≥ 4.96 mmol/L).

    II. Hepatic: Total bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 3 in patients with liver metastases or know history of Gilbert's disease); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times ULN (≤ 5 in patients with liver metastases); international normalized ratio (INR) < 1.5.

    III. Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 40 mL/min/1.73 m2 based on Cockcroft-Gault glomerular filtration rate estimation for patients with creatinine levels above institutional normal.
17. Resolution of all acute toxic effects of prior anti-cancer therapy to grade ≤ 1 as determined by the US National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v.5.0) (except for alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
18. Women of childbearing potential (WOCBP) who are sexually active with a non-sterilized male partner must have a negative serum pregnancy test within 14 days before study treatment initiation. In addition, they must agree to use one highly effective method of birth control from the time of screening until 2 months after the last dose of study treatments. Female patients must refrain from egg cell donation and breastfeeding during this same period.

    Note: Due to a potential loss of effectiveness of hormonal contraceptives caused by interaction with study intervention, if WOCBP use hormonal contraceptives (including oral hormonal contraceptives), they must use either another form of non-hormonal highly effective contraception or a reliable barrier method.
19. Male participants who are sexually active with a WOCBP partner must be surgically sterile or using an acceptable method of contraception from the time of screening until 4 months after the last administration of the study drug. Male participants must not donate or bank sperm during this same period.
20. Patient must be accessible for treatment and follow-up.

Exclusion Criteria:

Any patient meeting ANY of the following criteria will be excluded from the study:

1. Major surgery within four weeks of the start of treatment.
2. Type I leptomeningeal disease per ESMO-EANO guidelines.
3. Have received prior radiotherapy within two weeks before the first dose of Study treatment (four weeks in case of radiation therapy of the central nervous system). Participants must have recovered from all radiation-related toxicities, not require steroids, and not have had radiation pneumonitis.
4. Treatment with approved or investigational cancer therapy within14 days prior to initiation of Study treatment.
5. Any of the following cardiac criteria:

   I. Mean resting corrected QT interval (ECG interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTc) > 470 msec obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value.

   II. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec).

   III. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval.
6. Clinically significant cardiovascular disease (either active or within 6 months prior to enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥ II), cerebrovascular accident or transient ischemic attack, symptomatic bradycardia, requirement for anti-arrhythmic medication. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2.
7. Known clinically significant active infections not controlled with systemic treatment (bacterial, fungal, viral including HIV positivity).
8. Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact on drug absorption.
9. Peripheral neuropathy grade ≥ 2.
10. History of extensive, disseminated, bilateral, or presence of NCI CTCAE grade 3 or 4 interstitial fibrosis or interstitial lung disease (ILD) including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, ILD, obliterative bronchiolitis, and pulmonary fibrosis. Patients with a history of prior radiation pneumonitis are not excluded.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise the protocol objectives in the opinion of the Investigator.
12. Presence or history of any other primary malignancy other than NSCLC within 5 years prior to enrollment into the study.

    Note: Patients with a history of adequately treated basal or squamous cell carcinoma of the skin or any adequately treated in situ carcinoma may be included in the study.
13. Current use or anticipated need for drugs that are known to be strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or inducers.

    Note: midazolam requires diligent monitoring in situations where there is an unprecedented necessity for co-administration. These cases should be discussed with the study's medical monitor.
14. Patients requiring concomitant use of chronic systemic (intravenously [IV] or oral) corticosteroids at doses higher than 8 mg dexamethasone per day or other immunosuppressive medications except for managing adverse events (AEs); (inhaled steroids or intra articular steroid injections are permitted in this study).

    Note: The use of stable corticosteroid therapy in patients with brain metastases should be discussed with the Sponsor's Medical Monitor.
15. Hypersensitivity to the Study drug or any of its ingredients.
16. Prior exposure to other investigational medical products within five times the half-life of the drug/metabolites before the Screening Visit.
17. Contraindications to MRI, including but not limited to claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective Response Rate (IC-ORR) | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of IC-ORR at any timepoint defined as the rate of patients with partial response (PR) or complete response (CR) for IC lesions, as determined locally by the investigator as judged by best CNS response according to the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) for intracranial (IC) lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of CBR, defined as the rate of patients with objective response (CR or PR), or stable disease (SD) for IC lesions for at least 24 weeks, as determined locally by the investigator using RANO-BM.
Disease Control Rate (DCR) for IC lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of DCR, defined as the percentage of patients with advanced cancer whose therapeutic intervention has led to a CR, PR, or SD for IC lesions, as determined locally by the investigator using RANO-BM.
Time to Response (TTR) for IC lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of TTR, defined as the period from the treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a CR or PR for IC lesions, as determined locally by the investigator using RANO-BM.
Duration of Response (DoR) for IC lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of DoR, defined as the period from the first occurrence of a documented objective response to disease progression or death from any cause, observed for patients who achieved a CR or PR for IC lesions, as determined locally by the investigator using RANO-BM.
Objective Response Rate for extracranial (EC) and overall lesions (EC-ORR) | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of EC-ORR at any timepoint defined as the rate of patients with partial response (PR) or complete response (CR) for EC and overall lesions, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v.1.1) criteria.
CBR for EC and overall lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of CBR at any timepoint defined as the rate of patients with objective response (CR or PR), or SD for EC and overall lesions, for at least 24 weeks, as determined locally by the investigator using RECIST v.1.1
DCR for EC and overall lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of DCR, defined as the percentage of patients with advanced cancer whose therapeutic intervention has led to a CR, PR, or SD for EC and overall lesions, as determined locally by the investigator using RECIST v.1.1
TTR for EC and overall lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of TTR, defined as the period from the treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a CR or PR for EC and overall lesions, as determined locally by the investigator using RECIST v.1.1
DoR for EC and overall lesions | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the efficacy in terms of DoR, defined as the period from the first occurrence of a documented objective response to disease progression or death from any cause, observed for patients who achieved a CR or PR for EC and overall lesions, as determined locally by the investigator using RECIST v.1.1.
Best percentage of change in tumor burden | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To evaluate the best percentage of change in tumor burden determined locally by the investigator using RANO-BM criteria for IC lesions and RECIST v.1.1 for EC and overall lesions.
Progression-Free Survival (PFS) | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the PFS, defined as the period from treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, determined locally per RANO-BM criteria for IC lesions and RECIST criteria v.1.1 for EC and overall lesions.
Overall Survival (OS) | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To determine the OS, defined as the period from treatment initiation to death from any cause, determined locally by the investigator.
Neurologic function | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To assess the patient neurologic function with the Neurologic Assessment in Neuro-Oncology (NANO) scale
Quality of life (QoL) with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-30) | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To evaluate changes from baseline and during repotrectinib treatment in terms of patient-reported outcome (PRO) assessments of QoL and treatment-related symptoms as measured by EORTC QLQ-C30 scale.
  EORTC QLQ-C30 scale aims to measure cancer patients' physical, psychological and social functions. Scale and single items are transformed into scores ranging from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
QoL with the brain cancer specific questionnaire (QLQ-C20). | From date of inclusion until the date of first documented progression or date of death from any cause or treatment discontinuation from any other reason, whichever came first, assessed through study completion, an average of 13 months.
  To evaluate changes during repotrectinib treatment in terms of PRO assessments of QoL and treatment-related symptoms as measured by EORTC QLQ-C20 scale.
  EORTC QLQ-BN20 brain specific tool aims to measure the effects of brain tumors and its treatment on symptoms, functions and health-related quality of life.
  Scale and single items are transformed into scores ranging from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Safety and tolerability | Through study completion, an average of 13 months.
  To evaluate the safety and toxicity profile of treatment with of repotrectinib as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

OTHER OUTCOMES:
Exploratory endpoint: Genetic studies using blood samples to investigate the potential association with clinical outcomes | Through study completion, an average of 13 months.
  Gene expression profiling analyses performed on blood samples to investigate the potential association with clinical outcomes.
Exploratory endpoint: ROS1 gene expression analysis using baseline tissue samples to investigate the potential association with clinical outcomes | Through study completion, an average of 13 months.
  ROS1 gene expression analysis performed on baseline tumor tissue samples to investigate the potential association with clinical outcomes.
Exploratory endpoint: Analysis of medical imaging to identify potential biomarkers associated with clinical outcomes | Through study completion, an average of 13 months.
  Analysis of oncological biomarkers, such as growth rate of tumor derived by tumor growth rate modeling or tumor heterogeneity according to quantitative estimation through radiomics, may be performed on radiological images to investigate the potential association with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Preusser, md, Principal Investigator — Medical University of Vienna, Vienna General Hospital (Austria); Barbara Kiesewetter, MD, Principal Investigator — Medical University of Vienna, Vienna General Hospital (Austria); Thorsten Füreder, MD, Principal Investigator — Medical University of Vienna, Vienna General Hospital (Austria)
Locations (15):
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Medical University of Vienna, Vienna
- Spain (13):
  - Hospital de Vinalopó, Elche, Alicante
  - UOMI Cancer Center, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Institut Català d' Oncologia Girona (ICO), Girona, Girona
  - Hospital Beata María Ana, Madrid, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario de León, León
  - Hospital Lucus Agusti, Lugo
  - Hospital Universitario Vithas Madrid La Milagrosa, Madrid
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Clínico Universitario de Valencia, Valencia